CLINICAL TRIAL: NCT02075164
Title: Unravelling the Pathogenetic Mechanisms of Fructose in Comparison to Glucose Consumption as Multiple Hit in the Pathogenesis and Progression of Non-alcoholic Fatty Liver Disease (NAFLD) - an Exploratory Trial
Brief Title: Unravelling Mechanisms of Fructose vs Glucose Consumption in the Pathogenesis and Progression of NAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Michael Trauner, MD (Other)
Collaborators: Wiener Wissenschafts-, Forschungs- und Technologiefonds (Unknown)
Responsible Party: Sponsor-Investigator, Prof. Michael Trauner, MD, Professor, MD, Head and Chair of the Division of Gastroenterology and Hepatology, Department of Internal Medicine III, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Fru2.0
Record Dates: First submitted 2014-02-06; First posted 2014-03-03 (Estimated); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Non-alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis
Keywords: Non-alcoholic Fatty Liver Disease; Non-alcoholic steatohepatitis; NAFLD; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Fructose; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fructose (Experimental): Volunteers will be challenged with oral 150g Fructose per day for 56 days.
  Interventions: Dietary Supplement: Fructose; Dietary Supplement: Glucose
- Glucose (Experimental): Volunteers will be challenged with oral 167g Fructose per day for 56 days.
  Interventions: Dietary Supplement: Fructose; Dietary Supplement: Glucose
- NAFLD (No Intervention): Patients with confirmed simple fatty liver will be compared at baseline with other arms.
- NASH (No Intervention): Patients with confirmed non-alcoholic steatohepatitis will be compared at baseline with other arms.

INTERVENTIONS:
Dietary Supplement: Fructose — High oral Fructose challenge (150g per day for 56 days)
  Arms: Fructose; Glucose
Dietary Supplement: Glucose — Dietary Supplement: High oral Fructose challenge (167g per day for 56 days)
  Arms: Fructose; Glucose

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) comprises a spectrum ranging from simple fatty liver over steatohepatitis (NASH) to liver cirrhosis and cancer (HCC) and is a major and increasing health problem affecting nearly 40% of the general population. Moreover, NAFLD is an important risk factor for progression of diabetes and atherosclerosis. However, the pathomechanisms determining disease progression are poorly understood. The overall aim of this project is to test the central hypothesis that excessive fructose consumption provides a multiple metabolic hit in the pathogenesis and progression of NAFLD/NASH by impairment of hepatic lipid homeostasis and mitochondrial function resulting in hepatic lipotoxicity with inflammasome activation and disturbed interorgan cross-talk among insulin sensitive tissues.

DETAILED DESCRIPTION:
To achieve these goals we will address the following specific hypotheses that

* Fructose-induced changes in lipid composition of hepatocellular stores determine lipotoxicity which may be associated with abnormalities in mitochondrial function, energy homeostasis, inflammasome activation and cellular injury in progression to NASH, effects which will be compared to glucose
* Non-invasive characterization of fructose (compared to glucose)-induced lipotoxic hepatic and extrahepatic metabolic risk profiles (lipid composition and energy metabolism) obtained by magnetic resonance spectroscopy (MRS) will identify patients with NASH
* Severity of fructose (compared to glucose)-induced lipotoxic lipid and adenosine triphosphate (ATP) derangements (identified by MRS) critically determines the degree of insulin resistance and abnormalities in hepatic glucose and lipid metabolism
* Compensatory hyperinsulinemia, secondary to skeletal muscle insulin resistance, may be a primary mechanism of hepatic lipotoxicity and progression to NASH
* Gender differences in the hepatic and systemic metabolic response to fructose are mediated by the impact of female sex hormones and their nuclear receptors on hepatic lipid metabolism, mitochondrial function and inflammasome activation.
* Age differences in the hepatic and systemic metabolic response to fructose are mediated by the impact of age related alterations on hepatic lipid metabolism and mitochondrial function.

These key hypotheses will be addressed by a translational research consortium including hepatologists, radiologists, physicists, endocrinologists and specialist in gender medicine allowing an integrated mechanistic approach to NAFLD. The strength of the current proposal comes directly from bridging basic science and clinical perspectives of different disciplines involved in the management of NAFLD, including cutting edge non-invasive technologies such as high field MRS metabolic profiling ('virtual metabolic liver biopsy') and mechanistic in vitro experiments. This project will provide novel mechanistic insights in the role of fructose as emerging hepatic 'toxin' in the pathogenesis and progression of NASH, as increasing health problem in Western society. Moreover, this study will clarify the impact of sex and gender on fructose-induced alterations in hepatic and systemic metabolism, providing a rational and scientific basis for future dietary interventions and regulatory actions.

ELIGIBILITY:
Inclusion criteria

1. Healthy men and women from 18 to 85, no disease history, no intake of regular medication, drugs, alcohol (alcohol consumption > 140 grams per week (or > 30g/day) 45) or herbals known to affect liver physiology, male and female (1:1), BMI <= 25.
2. Patients with prior confirmed (biopsy within 6 months prior to study) intrahepatic fat accumulation/simple fatty liver (NAFL), HbA1c < 6.5, male and female (1:1)
3. Patients with confirmed NASH (biopsy within 6 months prior to study), HbA1c < 6.5, male and female (1:1).
4. Signed informed consent, willing and able to perform study procedures.

General exclusion criteria (for all groups)

1. Pregnancy and lactation (blood/urine pregnancy test will be performed for female volunteers at baseline and week 4)
2. Imprisoned persons
3. Declined informed consent
4. Inflammatory bowel conditions (celiac disease, Crohn's disease, ulcerative colitis)
5. Prior bariatric surgery
6. Alcoholic steatohepatitis and/or alcohol consumption > 140 grams per week (or > 30g/day) 45
7. Other liver diseases (autoimmune, genetic, cholestatic, Wilson disease, Weber-Christian disease, partial lipodystrophy of the face sparing type, abetalipoproteinemia, and jejunal diverticulosis with bacterial overgrowth).
8. Virus hepatitis (A, B, C)
9. Known allergic reaction to the drugs used (see material and methods)
10. Intake of drugs known to accumulate intrahepatic lipids and significantly interfere with metabolism (e.g. steroids/glucocorticoids, tamoxifen, amiodarone, perhexiline maleate, antiretroviral agents, tetracycline, minocycline, certain pesticides) 45
11. Inability or contraindications to perform study procedures
12. Fructose malabsorption diagnosed by two consecutive positive fructose hydrogen breath test

MRI contraindications Study participants with claustrophobia Study participants carrying

* a cardiac pacemaker
* an insulin pump
* operation clips
* nerval stimulators
* implants or prostheses (e.g. ear implants, hip prostheses, heart valve, penile prosthesis)
* metal parts or metal fragments [e.g. metallic intrauterine devices (IUDs), marrow nail, metallic splinters or munition rests)
* metallic shunts or stents

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2013-05; Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Intrahepatic total fat and ipid composition assessed by Magnetic resonance spectroscopy | Healthy volunteers: Baseline, day 56 (8 weeks); NAFLD/NASH patients: Baseline
  At baseline and on the last day of the study (day 56) Magnetic resonance spectroscopy will be carried out in healthy volunteers. (Prior and after double-blinded fructose versus glucose consumption for 8 weeks in each healthy volunteer).
  In NAFLD and NASH patients Magnetic resonance spectroscopy will only be carried out at baseline, as this arms/groups do not undergo an oral fructose/glucose challenge.
  Baseline measures between healthy volunteers and NAFLD/NASH groups/arms will be compared to assess differences between healthy individuals and patients.
  Baseline and day 56 measures in healthy volunteers after fructose/glucose consumption will be compared to assess the influence of the dietary challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Trauner, Prof. MD, Principal Investigator — Division of Gastroenterology and Hepatology Department of Internal Medicine III Medical University of Vienna
Locations (1):
- Medical University of Vienna, General Hospital of Vienna Vienna, Vienna, Austria 1090, Vienna, Austria

REFERENCES:
- [Derived] Smajis S, Gajdosik M, Pfleger L, Traussnigg S, Kienbacher C, Halilbasic E, Ranzenberger-Haider T, Stangl A, Beiglbock H, Wolf P, Lamp T, Hofer A, Gastaldelli A, Barbieri C, Luger A, Trattnig S, Kautzky-Willer A, Krssak M, Trauner M, Krebs M. Metabolic effects of a prolonged, very-high-dose dietary fructose challenge in healthy subjects. Am J Clin Nutr. 2020 Feb 1;111(2):369-377. doi: 10.1093/ajcn/nqz271. PMID 31796953